CLINICAL TRIAL: NCT00188474
Title: A Prospective Study of Patient Centered Outcomes in the Management of Malignant Pleural Effusions
Brief Title: A Quality of Life Study re Management of Malignant Pleural Effusions
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 04-0233-CE
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Malignant Pleural Effusions
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: LCADLS, FACIT-PAL, FACIT-TS questionnaires — LCADLS, FACIT-PAL, FACIT-TS questionnaires

SUMMARY:
There is much data in the literature regarding optimal treatment approaches for malignant pleural effusions as assessed by patient outcomes. However, data on quality of life and satisfaction with treatment from the patient's perspective is not available.

DETAILED DESCRIPTION:
This study will compare various treatment strategies in the management of malignant pleural effusions with respect to:

1. Primary endpoint: the successful palliation of symptomatic pleural effusions as assessed by the London Chest Activity of Daily Living Scale (LCADLS)
2. Secondary endpoints:

   i) impact of treatment on patient quality of life as assessed by the Functional Assessment of Chronic Illness Therapy - Palliative patient (FACIT-PAL) questionnaire ii) Assessment of patient satisfaction with treatment received via Functional Assessment of Chronic Illness Therapy-Treatment Satisfaction (FACIT-TS) questionnaire iii)Pleurodesis success rates assessed by 2 and 6-week effusion control rates on CXR iv) Requirement of further hospitalizations or procedures for the treatment of recurrent effusions v) Comparison of morbidity and mortality rates for differing treatment approaches vi) comparison of cost in a Canadian health care setting for differing treatment approaches

ELIGIBILITY:
Inclusion Criteria:

* symptomatic pleural effusion
* history of malignant disease
* age greater that 18 years
* consent to participate in study

Exclusion Criteria:

* significant ipsilateral endobronchial disease
* prior ipsilateral, intra-pleural therapy, as defined by: prior chest tube placement for effusion, prior attempt at chemical/surgical pleurodesis, prior surgical pleurectomy
* active pulmonary or pleural infection
* granulocytes < 1500/mm3, platelets < 50,000/mm3
* systemic chemotherapy within 2 weeks
* allergy to talc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant pleural effusions
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2004-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
the successful palliation of symptomatic pleural effusions as assessed by the London Chest Activity of Daily Living Scale (LCADLS) | discharge, 2 wks and 6 wks

CONTACTS AND LOCATIONS:
Overall Officials: Gail Darling, MD, FRCS(C), Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - University Health Network, Toronto, Ontario
  - St. Joseph's Hospital, Toronto, Ontario